CLINICAL TRIAL: NCT01023464
Title: Tear Film Break-Up Time Evaluation of FID 114657
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-030
Record Dates: First submitted 2009-11-25; First posted 2009-12-02 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: tear film break-up time
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricants; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 (Other): FID 114657 or SootheXP
  Interventions: Other: FID114657; Other: SootheXP Emollient (Lubricant) Eye Drops
- Period 2 (Other): FID 114657 or SootheXP
  Interventions: Other: FID114657; Other: SootheXP Emollient (Lubricant) Eye Drops

INTERVENTIONS:
Other: FID114657 — artificial tears
Other: SootheXP Emollient (Lubricant) Eye Drops — artificial tears

SUMMARY:
To evaluate the effects of FID 114657 on tear film break-up time in dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent document and HIPAA privacy document must be read, signed and dated by the patient or legally authorized representative before conducting any procedures.
2. Patients (minimum age 18) with dry eye. Criteria for the diagnosis must include the following characteristics at Visit 1 (Screening): Patients' self-assessment of dry eye status (answer of at least Some of the time to the question, "How often have your eyes felt dry enough to want to use eye drops?");TFBUT <5 seconds in at least one eye; > Grade 1 for Meibomian Gland Expression in both eyes; Evidence of missing meibomian glands in both eyes.
3. Able and willing to follow study instructions.
4. Patients must have best-corrected visual acuity of 0.6 logMAR or better in each eye as assessed using an ETDRS chart at Visit 1.
5. Patients must not have used any topical ocular drops for approximately 24 hours prior to Visit 1.

Exclusion Criteria:

1. History or evidence of ocular or intraocular surgery in either eye within the past six months.
2. History or evidence of serious ocular trauma in either eye within the past six months.
3. Current punctal occlusion of any type (e.g., collagen plugs, silicone plugs).
4. History of intolerance or hypersensitivity to any component of the study medications.
5. History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia; active or recent varicella viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye.
6. Use of any concomitant topical ocular medications during the study period.
7. Patients using systemic medications that may contribute to dry eye (e.g. cold and allergy medications, tricyclic antidepressants, hormone replacement therapies) may not be enrolled in the study unless they have been on a stable dosing regimen for a minimum of 30 days prior to Visit 1. In addition, the dosing regimen must remain stable throughout the study.
8. Ocular conditions such as conjunctival infections, iritis, or any other ocular condition that may preclude safe administration of the test article.
9. Individuals unwilling to discontinue contact lens wear during the study period. Contact lens wear must have been discontinued at least one week prior to Visit 1.
10. Enrollment of investigator's office staff, relatives, or members of their respective households; or enrollment of more than one member of the same household.
11. Participation in an investigational drug or device study within 30 days of entering this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
tear film break-up time (TFBUT) | Instill assigned test article to both eyes and begin timing the evaluation process. Measure TFBUT at 15, 30, 60 and 120 minutes post instillation.

SECONDARY OUTCOMES:
Acute comfort | Immediately post instillation of test article

REFERENCES:
- [Result] Benelli U. Systane lubricant eye drops in the management of ocular dryness. Clin Ophthalmol. 2011;5:783-90. doi: 10.2147/OPTH.S13773. Epub 2011 Jun 10. PMID 21750611